CLINICAL TRIAL: NCT06694428
Title: Evaluation of Software for Interpreting Virological Results Indicated for the Diagnosis of Cytomegalovirus (CMV) Infection During Pregnancy and Intended for Health Professionals
Acronym: MyCMV
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240966
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Cytomegalovirus Infections; Maternal Primary Cytomegalovirus Infection
Keywords: Congenital cytomegalovirus (cCMV) infection; Maternal primary cytomegalovirus infection; Maternal Screening and Diagnosis; Decision-making algorithm
MeSH Terms: conditions — Cytomegalovirus Infections; Infections; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Pregnant women with prescription of a CMV serology including the search for CMV IgG and IgM antibodies, care at the Necker-Enfants Malades or Paul Brousse hospitals, with positive CMV IgM antibodies or in the grey zone of the technique and for whom the date of start of pregnancy is known.
  Interventions: Other: Reinterpretation of CMV serology results using the MyCMV tool on the basis of the serology results performed

INTERVENTIONS:
Other: Reinterpretation of CMV serology results using the MyCMV tool on the basis of the serology results performed — The CMV serology results of the patients will have been previously interpreted as part of the care on the basis of the entire virological file according to the reference method.
  These results will be reinterpreted using the MyCMV tool on the basis of the serology results performed (IgM, IgG, avidity), CMV PCR, the date of sampling and the date of the start of pregnancy (or last period). This reinterpretation by the tool will be carried out as part of the study and will not be communicated to the patient or to the doctor prescribing the virological analyses.

SUMMARY:
Congenital cytomegalovirus (CMV) infection is the most common congenital infection with a birth prevalence of 0.4% in Europe. It is the leading non-genetic cause of sensorineural hearing loss and a major cause of neurodevelopmental disabilities. The risk of intrauterine transmission is highest when primary infection occurs during pregnancy. Primary CMV infection is asymptomatic or causes non-specific symptoms and only serology can diagnose it with certainty.

The diagnosis of CMV infection is based on the combination of 2 or 3 serological markers and the interpretation of the results is more complex than for other infections and may require additional analyses and sometimes delay the diagnosis and the implementation of secondary prevention of CMV transmission to the fetus by the administration of valaciclovir. Indeed, the effectiveness of secondary prevention is conditioned by the early administration of treatment after the maternal primary infection.

The National Reference Center for Congenital CMV Infections at Necker Hospital, in collaboration with the virology laboratory at Paul Brousse Hospital, has developed the MyCMV "expert" tool, which is a decision-making algorithm that allows the interpretation of CMV serology and CMV PCR results.

The hypothesis of the study is that the use and provision of this MyCMV "expert" tool to health professionals (biologists, midwives and obstetricians) for the interpretation of virological results could avoid a delay in diagnosis and would allow patients to be referred more quickly to a prenatal diagnosis center for appropriate management of CMV infection.

The aim of the study is to evaluate the rate of detection of primary CMV infection in the first trimester of pregnancy using the MyCMV tool compared with the reference method (results interpreted by the centre's expert investigator).

DETAILED DESCRIPTION:
Congenital cytomegalovirus (CMV) infection is the most common congenital infection with a birth prevalence of 0.4% in Europe. It is the leading non-genetic cause of sensorineural hearing loss and a major cause of neurodevelopmental disabilities. The risk of intrauterine transmission is highest when primary infection occurs during pregnancy. Primary CMV infection is asymptomatic or causes non-specific symptoms and only serology can diagnose it with certainty.

The diagnosis of CMV infection is based on the combination of 2 or 3 serological markers and the interpretation of the results is more complex than for other infections and may require additional analyses and sometimes delay the diagnosis and the implementation of secondary prevention of CMV transmission to the fetus by the administration of valaciclovir. Indeed, the effectiveness of secondary prevention is conditioned by the early administration of treatment after the maternal primary infection.

The National Reference Center for Congenital CMV Infections at Necker Hospital, in collaboration with the virology laboratory at Paul Brousse Hospital, has developed the MyCMV "expert" tool, which is a decision-making algorithm that allows the interpretation of CMV serology and CMV PCR results.

The hypothesis of the study is that the use and provision of this MyCMV "expert" tool to health professionals (biologists, midwives and obstetricians) for the interpretation of virological results could avoid a delay in diagnosis and would allow patients to be referred more quickly to a prenatal diagnosis center for appropriate management of CMV infection.

The aim of the study is to evaluate the rate of detection of primary CMV infection in the first trimester of pregnancy using the MyCMV tool compared with the reference method (results interpreted by the centre's expert investigator). We also aim to evaluate the dating of the maternal primary infection in weeks of amenorrhoea and additional tests given by the MyCMV tool compared with the reference method.

For the study, the medical information of patients for whom CMV serology including the search for CMV IgG and IgM antibodies is prescribed in the Necker-Enfants Malades or Paul Brousse hospitals, with positive CMV IgM antibodies or in the grey zone of the technique and for whom the date of start of pregnancy is known, will be reinterpreted with the MyCMV tool without consequences on the care of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman
* And for whom a CMV serology including the search for CMV IgG and IgM antibodies is prescribed at the Necker-Enfants Malades or Paul Brousse hospital
* And with positive anti-CMV IgM or in the grey zone of the technique
* And for whom the date of start of pregnancy is known
* And who does not object to the use of their data in the context of this research

Exclusion Criteria: NA

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women.
Study Population: Pregnant women with prescription of a CMV serology including the search for CMV IgG and IgM antibodies, care at the Necker-Enfants Malades or Paul Brousse hospitals, with positive CMV IgM antibodies or in the grey zone of the technique and for whom the date of start of pregnancy is known.
Sampling Method: Non-Probability Sample
Enrollment: 491 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-04-04 (Estimated); Study Completion 2026-04-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the detection rate of primary CMV infection in the first trimester of pregnancy using the MyCMV tool | Time 0
  Detection of primary CMV infection in the first trimester of pregnancy by the MyCMV tool or by the reference method.
  In the context of this study, the reference method is the interpretation of the results by the expert investigator of the center, without using the MyCMV tool.

SECONDARY OUTCOMES:
Dating in weeks of amenorrhea of the date of primary infection by the MyCMV tool and by the reference method | Time 0
  Dating in weeks of amenorrhea of the date of primary infection by the MyCMV tool and by the reference method.
  In case of seroconversion of IgG or the presence of isolated IgM (followed by seroconversion in a subsequent serum) in the patient's previous results, evaluation of the dating in weeks of amenorrhea given by the MyCMV tool compared to the dating obtained by the reference method.
Recommendations for the conduct to be adopted for carrying out additional analysis by the MyCMV tool | Time 0
  Among the cases where it is not possible to conclude as to the occurrence of a primary infection during pregnancy on the basis of the available results, identification of the course of action to be taken for carrying out the additional analysis (on a previous sample, the same sample or a new sample) proposed by the reference method and the MyCMV tool.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Leruez-Ville, M.D., PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Jacques Fourgeaud, Pharma.D., PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: No